CLINICAL TRIAL: NCT05638854
Title: A Phase 1, 2-Part, Single Ascending Dose (SAD) Study to Evaluate the Safety and Pharmacokinetics (PK) of ZB002 in Healthy Volunteers (HVs) and Multiple Ascending Dose (MAD) Study to Evaluate the Safety and PK of ZB002 in Participants With Rheumatoid Arthritis (RA)
Brief Title: A Study to Evaluate Safety and Pharmacokinetics of ZB002 in Healthy Participants and Participants With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zenas BioPharma (USA), LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZB002-01-001
Record Dates: First submitted 2022-11-15; First posted 2022-12-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers; Rheumatoid Arthritis
Keywords: Healthy Volunteers; Healthy Subjects; Healthy Participants; Patients; Rheumatoid Arthritis; RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: SAD in Healthy Volunteers (Experimental): Healthy volunteers will receive a single dose of ZB002 or placebo
  Interventions: Drug: ZB002; Drug: Placebo
- Part B: MAD in RA Participants (Experimental): RA participants will receive ZB002 or placebo every 4 weeks (Q4W) × 3 administrations
  Interventions: Drug: ZB002; Drug: Placebo

INTERVENTIONS:
Drug: ZB002 — ZB002 will be administered subcutaneously as per schedule specified in the respective arm.
  Arms: Part A: SAD in Healthy Volunteers
Drug: Placebo — Placebo will be administered subcutaneously as per schedule specified in the respective arm.
  Arms: Part A: SAD in Healthy Volunteers
Drug: ZB002 — ZB002 will be administered subcutaneously as per schedule specified in the respective arm.
  Arms: Part B: MAD in RA Participants
Drug: Placebo — Placebo will be administered subcutaneously as per schedule specified in the respective arm.
  Arms: Part B: MAD in RA Participants

SUMMARY:
This double-blind, randomized, placebo-controlled study will assess the safety and pharmacokinetics of ZB002 in healthy participants and in participants with rheumatoid arthritis (RA). The study consists of 2 parts. Part A: Single Ascending Dose (SAD), which will include only healthy volunteers. Part B: Multiple Ascending Dose (MAD), will commence after completion of the SAD study and will include RA participants.

DETAILED DESCRIPTION:
Part A (SAD): Up to approximately 48 healthy volunteers across 6 cohorts randomized to receive ZB002 or placebo as a single dose.

Part B (MAD): Up to approximately 24 participants with RA across 3 cohorts randomized to receive ZB002 or placebo as multiple doses.

ELIGIBILITY:
Main Inclusion Criteria

Part A SAD (HV):

* Healthy male or female participants 18 to 55 years of age.
* Body weight ≥ 50 kg for male participants and ≥ 45 kg for female participants; body mass index of 18 to 35 kg/m^2 for both male and female participants.
* Considered in good health as determined by the Investigator.
* Female participants of child-bearing potential must agree to abstinence or use an effective form of contraception.
* Male participants must be surgically sterile or agree to use effective contraception.
* Willing and able to understand the characteristics and purposes of the study, including possible risks involved, and willing to comply with all the study requirements and provide written informed consent for the study.

Part B MAD (RA Participants):

* Male or female participants 18 to 70 years (inclusive) of age at Screening.
* Body mass index of ≥ 18.0 and ≤ 40.0 kg/m2.
* Diagnosis of RA and meeting the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism classification criteria for RA ≥ 3 months before Screening.
* Use of methotrexate at 7.5 to 25 mg/week for ≥ 3 months, with stable dosing for ≥ 4 weeks, before randomization. Hydroxychloroquine/chloroquine and/or sulfasalazine are allowed if started ≥ 3 months before randomization and a stable dose is maintained after the Screening Visit.

Main Exclusion Criteria

Part A SAD (HV):

* Surgery within 4 weeks before Screening or planned surgery during the clinical study.
* Use of prescription medications, biological products, or other medicines within 2 weeks before Study Day 1 or 5 half-lives of the product, whichever is greater. Use of over-the-counter medications or vitamins/dietary supplements within 7 days of dosing unless considered by the Investigator to not pose a risk or impact the study results.
* Treatment with any investigational drug within 30 days or 5 half-lives, whichever is greater, before the first dose of the study drug, or currently enrolled in another clinical study.
* Clinically significant ECG abnormality.
* Positive for HIV infection, active hepatitis C, or hepatitis B.
* Positive for COVID-19 virus.
* Positive QuantiFERON®-TB Gold or T-SPOT® test for Mycobacterium tuberculosis.
* Bacteria, viruses, systemic fungi, parasites, or other opportunistic infections within 30 days before Study Day 1.
* Documented history of drug abuse in the previous 12 months before Screening, or positive for urine drug screen on Screening and/or Day -1.
* Donated blood (including component blood) or lost > 400 mL within 3 months before Screening or received a transfusion within 3 months of Screening.
* History of relevant allergies (including allergy to any murine or human-derived protein or immunoglobulin products, rubber or latex, or other allergies that in the opinion of the Investigator make inclusion in the study inappropriate).
* Average daily smoking > 10 cigarettes or cigarette equivalents per day within 6 months of Screening.
* Consume > 14 standard units of alcohol per week (1 standard unit is equivalent to approximately 360 mL of beer, 45 mL of spirits with 40% alcohol, or 150 mL of wine) or a positive alcohol breath test on Day -1.

Part B MAD (RA Participants):

* Inflammatory joint disease other than RA. Note: Current diagnosis of secondary Sjogren's Syndrome is permitted.
* Surgery within 4 weeks before Screening or planned surgery during the clinical study.
* History of any malignancy within 5 years, except for successfully treated nonmelanoma skin cancer or localized carcinoma in situ of the cervix.
* Documented history of drug abuse in the previous 12 months before Screening (Days -28 to -1), or positive for urine drug screen for nonprescribed drugs other than cannabinoid at Screening.
* Any condition considered by the investigator to make participation in the study inappropriate.
* Donated blood (including component blood) or lost > 400 mL within 1 month before Screening or received a transfusion within 3 months of Screening.
* After the Screening Visit, corticosteroid use > 10 mg/day (prednisone equivalent) or increase in dose
* Positive for HIV infection, active hepatitis C, or hepatitis B.
* Test positive for Mycobacterium tuberculosis.
* Bacterial, viral, systemic fungal, parasitic, or opportunistic infection not resolved at least 14 days before Study Day 1 or expected to be treated with antibiotics during the Treatment Period, or history of recurrent infections.
* Employees or related personnel of the study site, the sponsor, or contract research organization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability in HVs | Day 1 through Day 120
  To evaluate the safety and tolerability of ZB002 in HVs by assessing the number, severity and type of adverse events, including changes in laboratory safety test and electrocardiogram (ECG)
Part B: Safety and Tolerability of multiple doses of ZB002 in participants with RA | Day 1 through Day 176
  To evaluate the safety and tolerability of ZB002 in participants with RA by assessing the number of participants with Treatment-emergent adverse events (TEAEs), serious TEAEs, and TEAE leading to discontinuation

SECONDARY OUTCOMES:
Part A: Maximum observed serum concentration (Cmax) | Day 1 through Day 120
  Pharmacokinetics
Part A: Time for Cmax (Tmax) | Day 1 through Day 120
  Pharmacokinetics
Part A: Area under the concentration-time curve from time zero extrapolated to infinity (AUCinf) | Day 1 through Day 120
  Pharmacokinetics
Part A: AUC from time 0 to the last quantifiable concentration (AUClast) | Day 1 through Day 120
  Pharmacokinetics
Part A: Terminal half-life (t1/2) | Day 1 through Day 120
  Pharmacokinetics
Part A: Apparent clearance following extravascular dosing (CL/F) | Day 1 through Day 120
  Pharmacokinetics
Part A: Apparent volume of distribution following extravascular administration (Vz/F) | Day 1 through Day 120
  Pharmacokinetics
Part B (All Doses): Serum trough concentration (Ctrough) | Day 1 through Day 176
  Before repeat-dose administration (or at the end of the dosing interval [tau] after the final dose)
Part B (Doses 1 and 3): Maximum observed serum concentration (Cmax) | Day 1 through Day 176
  Pharmacokinetics
Part B (Doses 1 and 3): Time for Cmax (Tmax) | Day 1 through Day 176
  Pharmacokinetics
Part B (Doses 1 and 3): AUC over the dosing interval, tau (AUCtau) | Day 1 through Day 176
  Pharmacokinetics
Part B (Doses 1 and 3): Accumulation ratio of Cmax (ARCmax) | Day 1 through Day 176
  Pharmacokinetics
Part B (Doses 1 and 3): Accumulation ratio of AUC (ARAUC) | Day 1 through Day 176
  Pharmacokinetics
Part B (Dose 3 only): Area under the concentration-time curve from time zero extrapolated to infinity (AUCinf) | Day 1 through Day 176
  Pharmacokinetics
Part B (Dose 3 only): Terminal half-life (t1/2) | Day 1 through Day 176
  Pharmacokinetics
Part B (Dose 3 only): AUC from time 0 to the last quantifiable concentration (AUClast) | Day 1 through Day 176
  Pharmacokinetics
Part B (Dose 3 only): Apparent clearance following extravascular dosing (CL/F) | Day 1 through Day 176
  Pharmacokinetics
Part B (Dose 3 only): Apparent volume of distribution following extravascular (Vz/F) | Day 1 through Day 176
  Pharmacokinetics
Part B: Serum anti-ZB002 antibody prevalence and incidence | Day 1 through Day 176
Part B: Cytokine/chemokine secretion in ex vivo stimulated whole blood | Day 1 through Day 176
  Pharmacodynamic

CONTACTS AND LOCATIONS:
Locations (2):
- Veritus Research, Melbourne, Australia
- NZCR New Zealand Clinical Research, Christchurch, New Zealand